CLINICAL TRIAL: NCT04667169
Title: Comparison of Post-operative Bleeding Incidence in Laser Haemorrhoidoplasty Versus Laser Haemorrhoidoplasty With Haemorrhoidal Artery Ligation: A Double-Blinded Randomized Controlled Trial
Brief Title: Bleeding in Laser Haemorrhoidoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Lim Shu Yu, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMRR-15-1112-24065
Record Dates: First submitted 2020-11-26; First posted 2020-12-14 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Hemorrhoids
Keywords: Laser Haemorrhoidoplasty; Haemorrhoidal Artery Ligation; Haemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Haemorrhoidoplasty (Experimental): A stab incision was made at the ano-cutaneous junction and the anodermis was tunneled with artery forceps to the pedicle of the haemorrhoids. The laser catheter was introduced submucosally towards the pedicle guided by a visible beam to ascertain the exact location of the laser fibre. This was then followed by about six pulsed laser energy delivered at five mm interval, while gradually withdrawing the laser catheter.
  Interventions: Procedure: Laser Haemorrhoidoplasty
- Haemorrhoidal Artery Ligation (Experimental): In addition to the delivery of laser energy as per the procedure described above, each identified pedicle was ligated with a suture, without Doppler guidance.
  Interventions: Procedure: Haemorrhoidal Artery Ligation

INTERVENTIONS:
Procedure: Haemorrhoidal Artery Ligation — Post-operatively, all subjects were given tablet Paracetamol 1 gm six hourly and Capsule Celecoxib 200 mg 12 hourly as pain control for five days. They were given Syrup Lactulose 15 cc 12 hourly for one week to prevent constipation. Subjects were discharged on the same day or one day after surgery. All patients were assessed in the clinic by a nurse/medical officer blinded to the type of procedure performed on post-operative 24 hours, one week and six weeks.
  Arms: Haemorrhoidal Artery Ligation
Procedure: Laser Haemorrhoidoplasty — Post-operatively, all subjects were given tablet Paracetamol 1 gm six hourly and Capsule Celecoxib 200 mg 12 hourly as pain control for five days. They were given Syrup Lactulose 15 cc 12 hourly for one week to prevent constipation. Subjects were discharged on the same day or one day after surgery. All patients were assessed in the clinic by a nurse/medical officer blinded to the type of procedure performed on post-operative 24 hours, one week and six weeks.
  Arms: Laser Haemorrhoidoplasty

SUMMARY:
Treatment options for haemorrhoid can be classified mainly into lifestyle modification, medical and procedural. Laser haemorrhoidoplasty (LHP) is a minimally invasive procedure which is effective in treating grade 2-4 haemorrhoids. However, one of the significant complications is post-operative bleeding. Some surgeons supplemented haemorrhoidal artery ligation (HAL) to help minimize post-operative bleeding, however, its effectiveness has not been formally evaluated. This study aims to compare the effectiveness of supplementation of HAL to LHP in reducing the incidence of post-operative bleeding. It was hypothesize that supplementation of HAL to LHP is not effective in reducing the post-operative bleeding incidence and is unnecessary. The study was designed as a double-blind, randomized controlled trial involving 78 patients who underwent laser haemorrhoidoplasty in Universiti Malaya Medical Centre, Malaysia from November 2016 to October 2018. The study compared the post-operative bleeding incidence of laser haemorrhoidoplasty (LHP) only (n=38) versus laser haemorrhoidoplasty with haemorrhoidal artery ligation (LHP + HAL) (n=38). Assessment of bleeding using verbal rating scale (VRS) and Clavien-Dindo score is made at post-operative 24 hours, one week and six weeks. Pain score, the presence of perianal swelling and operation time were documented.

DETAILED DESCRIPTION:
Symptomatic haemorrhoids is a very common condition. The exact number of haemorrhoid sufferers is difficult to estimate because many do not seek medical help and rely on over the counter medications. Treatment options for haemorrhoids can be largely classified into lifestyle modification, medical and procedural. Procedural treatment can be further classified into excisional (involves excision of tissue) and non-excisional. Many procedures have been described and there is a preference for minimally invasive procedures and to avoid excisional procedures currently as they cause significantly more pain. Furthermore, many studies have shown that the post-operative complication rates and recurrence rates are relatively low for non-excisional procedures. In recent years, LHP had been introduced. It is an example of non-excisonal procedure for haemorrhoid. The delivery of laser energy to the anal cushion results in inflammation and scarring, which leads to contraction and fixation of haemorrhoids. The potential advantage of this procedure is less pain, as it does not involve. excision or passage of suture. Nevertheless, one of the post-operative conditions observed after LHP is bleeding. As this is a rather new procedure, there are limited studies conducted and the incidence of post-operative bleeding for laser haemorrhoidoplasty is not reported. To overcome this, some surgeons supplement haemorrhoidal artery ligation to laser haemorrhoidoplasty to minimize the incidence of post-operative bleeding, of which its effectiveness has not been formally evaluated. Moreover, the reported incidence of post-operative bleeding for HAL is 19-22%. In our institution experience, the post-operative bleeding rate for LHP is 1-2%. Therefore, the investigators hypothesize that supplementation of HAL to LHP is not effective in reducing the post-operative bleeding incidence and is unnecessary. This is an interventional study and is designed as a double-blinded randomized controlled trial to look into the post-operative bleeding incidence of patients undergoing LHP only versus LHP + HAL in UMMC. The study commenced in November 2016 and completed recruitment in October 2018. To show the effectiveness of supplementation of HAL to LHP in reducing the post-operative bleeding incidence, the investigators needed to study 35 experimental subjects and 35 control subjects to be able to reject the null hypothesis that the failure rate for experimental and control subjects are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05. When a 10% dropout rate was factored in, the investigators needed 38 subjects in each arm. The investigators will use an uncorrected chi-squared statistic to evaluate this null hypothesis. Randomization in blocks of four was used to assign the LHP only group and LHP + HAL group. Each procedure after randomized was placed in an individually numbered envelope. Prior to the start of operation, the operating surgeon randomly selects one envelop. All patients had general anaesthesia or regional anaesthesia. A standard dose of Intravenous Cefoperazone 2 gm and Intravenous Metronidazole 500 mg was given. Post-operatively, all subjects were given tablet Paracetamol 1 gm six hourly and Capsule Celecoxib 200 mg 12 hourly as pain control for five days. They were given Syrup Lactulose 15 cc 12 hourly for one week to prevent constipation. Subjects were discharged on the same day or one day after surgery. All patients were assessed in the clinic by a nurse/medical officer blinded to the type of procedure performed on post-operative 24 hours, one week and six weeks. There were a total of 76 patients recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above
* Diagnosed with symptomatic haemorrhoid
* Able to give informed consent
* Fit to undergo anaesthesia
* Agreeable for randomization and shows no preference for either group

Exclusion Criteria:

* Have stated a preference toward a certain treatment option
* Haemorrhoid condition requiring emergency surgery
* Haemorrhoids condition associated with other anorectal pathology such as fistula in ano, perianal abcess, and anal fissure
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Overall post-operative bleeding incidence | One day
  The assessment was made using of bleeding using verbal rating scale and Clavien-Dindo score.
Overall post-operative bleeding incidence | One week
  The assessment was made using of bleeding using verbal rating scale and Clavien-Dindo score.
Overall post-operative bleeding incidence | Six weeks
  The assessment was made using of bleeding using verbal rating scale and Clavien-Dindo score.

SECONDARY OUTCOMES:
Pain score | One day
  The assessment was made using the visual analogue scale (VAS)
Pain score | One week
  The assessment was made using the visual analogue scale (VAS)
Pain score | Six weeks
  The assessment was made using the visual analogue scale (VAS)
The presence of perianal swelling | One day
  The assessment was documented as its presence or the absence
The presence of perianal swelling | One week
  The assessment was documented as its presence or the absence
The presence of perianal swelling | Six weeks
  The assessment was documented as its presence or the absence
Operation time | Day 0
  The assessment was made based on the clinical records

CONTACTS AND LOCATIONS:
Overall Officials: Shu Yu Lim, MSurg, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim SY, Rajandram R, Roslani AC. Comparison of post-operative bleeding incidence in laser hemorrhoidoplasty with and without hemorrhoidal artery ligation: a double-blinded randomized controlled trial. BMC Surg. 2022 Apr 21;22(1):146. doi: 10.1186/s12893-022-01594-z. PMID 35449097